CLINICAL TRIAL: NCT02207426
Title: A Phase 1 Study in Healthy Volunteers Investigating the Delivery of Tobramycin Using the TobrAir® 6.0 Device Compared With the Delivery of Marketed Tobramycin Nebuliser Solution (TOBI®) by PARI LC® PLUS and PARI TurboBoy® SX and With Delivery of Tobramycin by the TOBI® Podhaler™ Device, Using Pharmacokinetic and Pharmacoscintigraphic Methods.
Brief Title: Pharmacokinetic and Pharmacoscintigraphic Comparison of TobrAir® 6.0 With TOBI® and TOBI® Podhaler™
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmaero ApS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TobrAir - CT0040; 2013-005288-19 (EudraCT Number)
Record Dates: First submitted 2014-08-01; First posted 2014-08-04 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Healthy
Keywords: Healthy volunteers
MeSH Terms: interventions — Tobramycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- TobrAir® 6.0 (Experimental): Tobramycin 75mg inhalation solution
  Interventions: Drug: Tobramycin
- TOBI® / PARI LC® PLUS Nebulizer (Experimental): Tobramycin 300mg nebulizer solution
  Interventions: Drug: Tobramycin
- TOBI® Podhaler™ (Experimental): Tobramycin 112mg (4x28mg) inhalation powder
  Interventions: Drug: Tobramycin

INTERVENTIONS:
Drug: Tobramycin

SUMMARY:
This study compares pharmacokinetic profiles of tobramycin delivered by TobrAir® 6.0 device with TOBI® nebulizer system and the TOBI® Podhaler™ device. In addition, lung deposition of tobramycin delivered by TobrAir® 6.0 device and by TOBI® nebulizer system will be determined.

DETAILED DESCRIPTION:
This is an open-label, randomized, single dose, cross-over study in healthy subjects. Each subject receives tobramycin with 3 different inhalation devices:

* 75 mg tobramycin delivered to the airways via TobrAir® 6.0.
* 300 mg tobramycin (TOBI®) delivered to the airways via the PARI LC® PLUS/PARI TurboBoy® SX.
* 112 mg tobramycin (4x28mg dry powder capsules) delivered to the airways via the TOBI® Podhaler™.

Each dose is separated by a minimum washout of at least 68 h.

Blood samples for PK analysis of tobramycin will be collected at regular time intervals until 24 h post-dose. For TobrAir 6.0 and TOBI/PARI only, all dosed subjects will undergo scintigraphic assessments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or non-pregnant, non-lactating healthy females
* Aged 18 to 65 years
* Body mass index of 18.0 to 29.0 kg/m2 or, if outside the range, considered not clinically significant by the investigator
* Must provide written informed consent
* Must agree to use an adequate method of contraception

Exclusion Criteria:

* Participation in a clinical research study within the previous 3 months
* Subjects who have previously been enrolled in this study
* Females of childbearing potential who are pregnant or lactating (female subjects must have a negative urine pregnancy test at admission and be using an appropriate method of contraception)
* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study
* History of chronic respiratory disorders (including asthma) as judged by the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-07; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Bioavailability of tobramycin | 3 days
  Bioavailability of tobramycin

SECONDARY OUTCOMES:
Scintigraphic measurement of lung deposition of radiolabelled tobramycin | 1 day
  Scintigraphic measurement of lung deposition of radiolabelled tobramycin

CONTACTS AND LOCATIONS:
Overall Officials: Pharmaero ApS Pharmaero ApS, Study Director — Pharmaero ApS
Locations (1):
- Quotient Clinical, Nottingham, United Kingdom